CLINICAL TRIAL: NCT05000177
Title: Alterations in Corticospinal and Neuromuscular Control of Shoulder Complex in Office Workers With Non-specific Chronic Neck Pain
Brief Title: Alterations in Central Control of Shoulder Muscles in Office Workers With Non-specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: YM110059F
Record Dates: First submitted 2021-07-18; First posted 2021-08-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Non-specific Chronic Neck Pain; Office Workers; Transcranial Magnetic Stimulation; Neuromuscular Control
Keywords: Non-specific chronic neck pain; Transcranial magnetic Stimulation; Corticospinal system; Scapular kinematics; Scapular muscles activation
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group: Non-specific chronic neck pain group (Other): Subjects with non-specific chronic neck pain will be included to perform 30-minute computer typing task and assess neurophysiological measurements of scapular muscles, scapular kinematics and muscle activation.
  Interventions: Other: 30-minute computer typing task
- Control group: Healthy subjects group (Other): Healthy subjects will be included to compare the differences in neurophysiological measurements of scapular muscles, scapular kinematics and muscle activation between healthy subjects and subjects with non-specific chronic neck pain. Subjects in this group will received the same assessment as the NCNP group.
  Interventions: Other: 30-minute computer typing task
- Pilot study: Healthy subjects group (Other): Healthy subjects will be included to test reliability of single-pulse and paired-pulse TMS, including its associated neurophysiological measurements, and also to test reliability of Liberty electromagnetic tracing system and surface electromyography. Subjects in this group will received the same assessment as the NCNP group.
  Interventions: Other: 30-minute rest

INTERVENTIONS:
Other: 30-minute computer typing task — The subject sits in front of a computer screen and perform computer typing tasks for 30 minutes. The same computer table and chair were used for all subjects. The height of the table and screen, and the distance of the keyboard from the subject were adjusted according to their familiar and comfortable position.
  Arms: Control group: Healthy subjects group; Experimental group: Non-specific chronic neck pain group
Other: 30-minute rest — Rest for 30 minutes
  Arms: Pilot study: Healthy subjects group

SUMMARY:
Non-specific chronic neck pain (NCNP) is commonly seen in office workers. Individuals with NCNP not only demonstrate impaired neck movement control and muscle activation, but also show abnormal scapular kinematics and muscle activation timing. Office workers with NCNP also show higher activity of upper trapezius during computer typing and have difficulty relaxing upper trapezius after typing. These changes related to scapula may increase strain over neck. In addition to the altered neuromuscular control, recent studies found neuroplasticity changes in the central nervous system on patients of chronic musculoskeletal disorders. Therefore, few studies found shifts and alterations of motor cortex representation of neck muscles in individuals with NCNP, which was correlated with delayed muscle activation of deep neck flexors muscle in functional activities. However, no studies have explored that whether this corticospinal adaptation also happens over scapular muscles, especially after a computer typing task. The objectives of this proposal are to investigate the differences in corticospinal and neuromuscular control of shoulder complex between office workers with and without NCNP. Thirty-five individuals with NCNP and 35 healthy controls will be recruited. Twenty young healthy subjects will be also recruited for a pilot study to test the reliability of all the measures. Scapular kinematics and muscle activation will be tested during arm elevation. Corticospinal parameters of trapezius and serratus anterior will be tested with transcranial magnetic stimulation (TMS), including active motor threshold, motor evoked potential, cortical silent period, short interval intracortical facilitation, short interval intracortical inhibition and cortical mapping. Corticospinal parameters, except cortical mapping, will be measured again after a 30-minute computer typing task. Scapular muscle activation will be also recorded during the typing task.

ELIGIBILITY:
Inclusion Criteria of Patients with Non-specific Chronic Neck Pain

1. Ages ranges from 20-40 years old
2. Work with the computer at least 25 hours per week
3. Neck pain of idiopathic origin ≥ 6 months during the past year
4. Minimum of 3/10 on the numerical rating scale (NRS) in past 7 days
5. No structural abnormalities which are confirmed by neck X-ray or negative results of all the following special tests

   * Exclude nerve root compression: Cervical distraction test and Spurling's test
   * Exclude cervical radiculopathy: Valsalva test
   * Exclude cervical instability: Alar ligament test and Sharp-Purser test
6. Specific head movements or maintaining the fixed posture for a long time reproduced neck pain

Inclusion Criteria of Healthy Subjects in the control group

1. Ages ranges from 20-40 years old
2. Work with the computer at least 25 hours per week
3. No history of neck and/or shoulder pain sustained over one week in the past one year

Inclusion Criteria of Healthy subjects in the Pilot Study

1. Ages ranges from 20-40 years old
2. No history of neck and/or shoulder pain sustained over one week in the past one year

Exclusion Criteria of Patients with Non-specific Chronic Neck Pain and All Healthy Subjects)

1. Any known pathology or impairment in the shoulder joint, which is the origin of neck pain
2. Current episode of neck pain related to a traumatic event (e.g., whiplash injury)
3. Have a history of cervical and/or shoulder pathology (e.g., fracture, dislocation, trauma, surgery of spinal or shoulder joint, inflammatory disease, frequent headache or dizziness)
4. Brain injury and neurological impairment (e.g., radiculopathy, myelopathy or stroke)
5. Systematic diseases (e.g., rheumatoid arthritis, ankylosing spondylitis), fibromyalgia, tumor
6. Contraindications to the use of transcranial magnetic stimulation (TMS), assessed with a safety screening questionnaire, including pregnancy, history of seizure, epilepsy and syncope, having cochlear implant, having medal implant and taking anti-depressant medication
7. Any kind of previous manual and/or movement therapy on upper extremity and neck during in recent 3 months

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Neurophysiological measures - Active motor threshold | Change from baseline AMT after 30-minute computer typing task or 30-minute rest
  Active motor threshold (AMT) will be described with the percentage (%) of maximum stimulator output (MSO).
Neurophysiological measures - Motor evoked potential | Change from baseline MEP after 30-minute computer typing task or 30-minute rest
  Motor evoked potential (MEP) will be described with millivolt (mV).
Neurophysiological measures - Cortical silent period | Change from baseline CSP after 30-minute computer typing task or 30-minute rest
  Cortical silent period (CSP) will be measured with millisecond (ms)
Neurophysiological measures - Short interval cortical inhibition | Change from baseline SICI after 30-minute computer typing task or 30-minute rest
  Short interval cortical inhibition (SICI) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is below 5 ms
Neurophysiological measures - Short interval cortical facilitation | Change from baseline SICF after 30-minute computer typing task or 30-minute rest
  Short interval cortical facilitation (SICF) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is above 5 ms
Neurophysiological measures - Area of cortical mapping | Before 30-minute computer typing task
  Area of cortical mapping will be described with square millimeter (mm2)
Neurophysiological measures - Volume of cortical mapping | Before 30-minute computer typing task
  Volume of cortical mapping will be calculated with multiplying summation of motor evoke potentials on the map (mV) by the area of the map (mm2) with the unit of mV*mm2
Neurophysiological measures - Center of gravity of cortical mapping | Before 30-minute computer typing task
  Center of gravity of cortical mapping will be described in a x-y coordinate system (mm).
Neurophysiological measures - Area of cortical mapping | Change from baseline area of cortical mapping after 30-minute rest (pilot subjects)
  Area of cortical mapping will be described with square millimeter (mm2)
Neurophysiological measures - Volume of cortical mapping | Change from baseline volume of cortical mapping after 30-minute rest (pilot subjects)
  Volume of cortical mapping will be calculated with multiplying summation of motor evoke potentials on the map (mV) by the area of the map (mm2) with the unit of mV*mm2
Neurophysiological measures - Center of gravity of cortical mapping | Change from baseline center of gravity of cortical mapping of cortical mapping after 30-minute rest (pilot subjects)
  Center of gravity of cortical mapping will be described in a x-y coordinate system (mm).

SECONDARY OUTCOMES:
Scapular kinematics during arm elevation | Before 30-minute computer typing task
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapula plane elevation at 30°, 60°, 90°, and 120°, and will be described with degree (°).
Scapular kinematics during performing the computer task | Change from baseline during the 30-minute computer typing task at 5, 10, 15, 20, 25, 30 minutes of the task
  The average of scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation will be calculated with a window of 10 seconds and will be described with degree (°).
Scapular muscles activation during arm elevation | Before 30-minute computer typing task
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, and serratus anterior will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°.
Scapular muscles activation during performing the computer task | Change from baseline during the 30-minute computer typing task at 5, 10, 15, 20, 25, 30 minutes of the task
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, and serratus anterior will be calculated with a window of 10 seconds and will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %).
Craniovertebral angle | Before 30-minute computer typing task
  Craniovertebral angle will be measured as the included angle between the tragus, C7 spinous process and the horizontal line and will be described with degree (°)
Craniovertebral angle | Change from baseline during the 30-minute computer typing task at 5, 10, 15, 20, 25, 30 minutes of the task
  Craniovertebral angle will be measured as the included angle between the tragus, C7 spinous process and the horizontal line and will be described with degree (°)
Scapular kinematics during arm elevation | Change from baseline scapular kinematics after 30-minute rest (pilot subjects)
  Scapular kinematics, including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapula plane elevation at 30°, 60°, 90°, and 120°, and will be described with degree (°).
Scapular muscles activation during arm elevation | Change from baseline scapular muscles activation after 30-minute rest (pilot subjects)
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, and serratus anterior will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°.
Craniovertebral angle | Change from baseline craniovertebral angle after 30-minute rest (pilot subjects)
  Craniovertebral angle will be measured as the included angle between the tragus, C7 spinous process and the horizontal line and will be described with degree (°)

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan